CLINICAL TRIAL: NCT00106639
Title: A 6-Month, Phase 2, Multicenter, Randomized, Open-Label, Comparative Study Of 2 Dose Levels Of CP-690,550 Administered Concomitantly With IL-2 Receptor Antagonist Induction Therapy, Mycophenolate Mofetil And Corticosteroids Versus A Tacrolimus-Based Immunosuppressive Regimen For The Prevention Of Allograft Rejection In De Novo Renal Allograft Recipients
Brief Title: A 6-Month Study Of CP-690,550 Versus Tacrolimus In Kidney Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A3921009
Record Dates: First submitted 2005-03-28; First posted 2005-03-29 (Estimated); Results first posted 2013-03-12 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-02

CONDITIONS: Kidney Transplantation
Keywords: tofacitinib; CP-690550; kidney transplant
MeSH Terms: interventions — tofacitinib; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CP-690,550 15 mg BID (Experimental)
  Interventions: Drug: CP-690,550
- CP-690,550 30 mg BID (Experimental)
  Interventions: Drug: CP-690,550
- tacrolimus (Active Comparator)
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Drug: CP-690,550 — 15 mg twice daily
  Arms: CP-690,550 15 mg BID
Drug: CP-690,550 — 30 mg twice daily
  Arms: CP-690,550 30 mg BID
Drug: tacrolimus — dose adjusted according to level
  Arms: tacrolimus

SUMMARY:
This Phase 2 study was designed to evaluate the safety and efficacy of 2 dose levels of CP-690,550 (15 mg twice daily and 30 mg twice) against tacrolimus, in combination with basiliximab induction, mycophenolate mofetil and corticosteroids, in kidney transplant patients. Stage 1 was to randomize approximately 54 subjects. After all Stage 1 subjects had completed 6 months of treatment, Stage 2 was to randomize an additional 195 subjects to the same treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a first-time kidney transplant
* Between the ages of 18 and 70 years, inclusive

Exclusion Criteria:

* Recipient of any non-kidney transplant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2005-05; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- United States (15):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Palo Alto, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Stanford, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Livingston, New Jersey
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Busque S, Leventhal J, Brennan DC, Steinberg S, Klintmalm G, Shah T, Mulgaonkar S, Bromberg JS, Vincenti F, Hariharan S, Slakey D, Peddi VR, Fisher RA, Lawendy N, Wang C, Chan G. Calcineurin-inhibitor-free immunosuppression based on the JAK inhibitor CP-690,550: a pilot study in de novo kidney allograft recipients. Am J Transplant. 2009 Aug;9(8):1936-45. doi: 10.1111/j.1600-6143.2009.02720.x. PMID 19660021
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921009&StudyName=A%206-Month%20Study%20Of%20CP-690%2C550%20Versus%20Tacrolimus%20In%20Kidney%20Transplant%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550 15 mg: CP-690,550 15 milligram (mg) tablet orally twice daily up to Month 6.
- CP-690,550 30 mg: CP-690,550 30 mg tablet orally twice daily up to Month 6.
- Tacrolimus: Tacrolimus 0.5 mg or 1 mg capsule administered orally as per local clinical practice up to Month 6.
Period: Overall Study
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Started | 20 | 20 | 21
Completed | 17 | 13 | 19
Not Completed | 3 | 7 | 2
Not completed — Adverse Event | 3 | 4 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Participant defaulted | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus | Total
Number analyzed (Participants) | 20 | 20 | 21 | 61
Age Continuous [Mean (Standard Deviation); unit: years] | 46.9 (8.5) | 44.3 (12.3) | 42.8 (11.8) | 44.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 4 | 8 | 24
  Male | 8 | 16 | 13 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Biopsy Proven Acute Rejection (BPAR) at Month 6
Description: BPAR categorized as acute rejection as interpreted by the central blinded pathologist according to the Banff 97 working classification.
Time Frame: Baseline up to Month 6
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
participants | 1 | 4 | 1

2. Primary Outcome: Glomerular Filtration Rate (GFR) by Nankivell Equation at Month 6
Description: GFR: index of kidney function described the flow rate of filtered fluid through the kidney. GFR was measured directly or estimated using established formulas. GFR was calculated by creatinine clearance (CLcr) using Nankivell equation. CLcr by Nankivell equation= (6.7 per serum creatinine) plus (0.25*body weight) minus (0.5*serum urea) minus (100 per square height) plus (35 for male/25 for female). A normal GFR is >90 milliliter/minute (mL/min), although children and older people usually have a lower GFR. Lower values indicated poor kidney function. A GFR <15 mL/min indicated kidney failure.
Time Frame: Month 6
Population: FAS included all randomized participants who received at least 1 dose of study medication. Here, N (Number of participants analyzed) signifies those participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 17 | 14 | 18
mL/min | 76.53 (10.04) | 71.50 (14.68) | 78.70 (12.61)

3. Secondary Outcome: Number of Participants With Treatment Failure
Description: Treatment failure was defined as the first occurrence of BPAR, graft loss, participant's death or premature discontinuation of study medication for any reason.
Time Frame: Month 3, 6
Population: FAS included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
participants
  Month 3 | 1 | 7 | 2
  Month 6 | 3 | 9 | 3

4. Secondary Outcome: Number of Participants With First Biopsy Proven Acute Rejection (BPAR) at Month 3
Description: as for outcome 1
Time Frame: Baseline up to Month 3
Population: FAS included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
participants | 0 | 4 | 1

5. Secondary Outcome: Number of Participants With First Biopsy Proven Chronic Allograft Nephropathy (BPCAN)
Description: BPCAN categorized as chronic allograft nephropathy as interpreted by the central blinded pathologist according to the Banff 97 working classification.
Time Frame: Month 3, 6
Population: FAS included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
participants
  Month 3 | 0 | 0 | 0
  Month 6 | 0 | 2 | 0

6. Secondary Outcome: Number of Participants With Ordered Categorical Severity of First Biopsy Proven Acute Rejection (BPAR)
Description: Ordered categorical severity of first BPAR was classified according to the Banff Classification. Grade IA: moderate tubulitis, grade IB: severe tubulitis, grade IIA: mild to moderate intimal arteritis, grade IIB: severe intimal arteritis, grade III: transmural arteritis. (Racusen et al: The Banff classification, 1999).
Time Frame: Month 3, 6
Population: FAS included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
participants
  Month 3: IA | 0 | 1 | 0
  Month 3: IB | 0 | 0 | 0
  Month 3: IIA | 0 | 2 | 0
  Month 3: IIB | 0 | 1 | 0
  Month 3: III | 0 | 0 | 0
  Month 6: IA | 0 | 1 | 0
  Month 6: IB | 0 | 0 | 0
  Month 6: IIA | 1 | 2 | 1
  Month 6: IIB | 0 | 1 | 0
  Month 6: III | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Ordered Categorical Severity of First Biopsy Proven Chronic Allograft Nephropathy (BPCAN)
Description: Ordered categorical severity of first BPCAN was classified according to the Banff Classification. Grade I: mild, grade II: moderate and grade III: severe interstitial fibrosis and tubular atrophy/loss. (Racusen et al: The Banff classification, 1999).
Time Frame: Month 3, 6
Population: FAS included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
participants
  Month 3: Any severity | 0 | 0 | 0
  Month 6: I | 0 | 2 | 0

8. Secondary Outcome: Number of Participants With Efficacy Failure
Description: Efficacy failure was the first occurrence of BPAR, graft loss or participant's death.
Time Frame: Month 3, 6
Population: FAS included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
participants
  Month 3 | 0 | 4 | 1
  Month 6 | 1 | 4 | 1

9. Secondary Outcome: Number of Participants With Graft Loss
Description: Graft loss was defined as graft nephrectomy, participant's death due to graft loss, re-transplantation, or return to dialysis for greater than or equal to (>=) 6 consecutive weeks.
Time Frame: Month 6
Population: FAS included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
participants | 0 | 0 | 0

10. Secondary Outcome: Number of Participants Who Died
Time Frame: Month 6
Population: FAS included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
participants | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Rejection
Description: Rejection was defined as first occurrence of BPAR, antibody mediated rejection, or suspicious for acute rejection.
Time Frame: Month 3, 6
Population: FAS included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
participants
  Month 3 | 1 | 4 | 1
  Month 6 | 2 | 4 | 1

12. Secondary Outcome: Population Pharmacokinetics (PK)
Description: Data for this Outcome Measure are not reported here because the analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the Participant Flow and Baseline Characteristics modules.
Time Frame: Pre-dose on Day 1, 3, 7, 14, Month 1, 3, 6, between 1 to 2 hours post-dose at Month 3 and between 3 to 4 hours post-dose at Month 6
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)

13. Secondary Outcome: Fluorescence-Activated Cell Sorting (FACS) of Lymphocyte Subsets
Description: The absolute cell counts of cluster of differentiation 8 (CD8): Cytotoxic T-lymphocytes reactive with major histocompatibility complex-1 (MHC-I), CD19: B- Lymphocytes, CD56: natural killer cells were determined using FACS, a specialized type of flow cytometry which sorts a heterogeneous mixture based upon the specific light scattering and fluorescent characteristics of each cell.
Time Frame: Baseline, Day 14, Month 1, 3, 6
Population: FAS included all randomized participants who received at least 1 dose of study medication. Here, N (Number of participants analyzed) signifies participants evaluable for this measure and 'n' signifies those participants evaluable at specific time points for each arm group respectively.
Measure: Mean (Standard Deviation); unit: cells per microliter (cells/mcL)
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 19 | 19 | 20
cells per microliter (cells/mcL)
  CD8: Baseline (n= 19, 19, 19) | 113.95 (80.91) | 114.05 (86.28) | 160.37 (146.56)
  CD8: Day 14 (n= 19, 19, 19) | 449.84 (327.09) | 471.79 (335.83) | 401.68 (313.64)
  CD8: Month 1 (n= 17, 18, 19) | 333.00 (226.24) | 354.39 (245.74) | 380.89 (257.68)
  CD8: Month 3 (n= 18, 18, 20) | 212.94 (133.54) | 252.72 (165.94) | 261.35 (156.93)
  CD8: Month 6 (n= 14, 11, 15) | 278.93 (198.35) | 201.09 (180.41) | 300.33 (195.51)
  CD19: Baseline (n= 19, 19, 19) | 69.74 (47.60) | 89.37 (74.13) | 111.32 (90.13)
  CD19: Day 14 (n= 19, 19, 19) | 353.68 (418.37) | 486.84 (410.32) | 303.95 (302.66)
  CD19: Month 1 (n= 17, 18, 19) | 282.41 (334.27) | 291.28 (208.87) | 343.58 (301.42)
  CD19: Month 3 (n= 18, 18, 20) | 128.39 (87.89) | 217.67 (276.83) | 168.20 (138.10)
  CD19: Month 6 (n= 14, 11, 15) | 156.50 (75.62) | 176.18 (169.09) | 188.80 (130.84)
  CD56: Baseline (n= 19, 19, 19) | 153.89 (120.10) | 127.84 (54.51) | 165.95 (97.05)
  CD56: Day 14 (n= 19, 19, 19) | 163.11 (162.67) | 151.68 (113.41) | 212.00 (294.38)
  CD56: Month 1 (n= 17, 18, 19) | 214.29 (399.94) | 101.11 (91.63) | 162.16 (80.31)
  CD56: Month 3 (n= 18, 18, 20) | 85.56 (69.64) | 70.00 (49.56) | 144.15 (80.96)
  CD56: Month 6 (n= 14, 11, 15) | 126.71 (153.23) | 36.27 (47.13) | 173.53 (119.79)

14. Secondary Outcome: Reticulocyte Count
Description: Reticulocytes are slightly immature red blood cells in the blood. Reticulocyte counts are reported as cells*10^3 per cubic millimeter (cells*10^3/mm^3).
Time Frame: Baseline, Day 14, Month 1, 3, 6
Population: FAS included all randomized participants who received at least 1 dose of study medication. Here 'n' signifies those participants evaluable at specific time points for each arm group respectively.
Measure: Mean (Standard Deviation); unit: cells*10^3/mm^3
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
cells*10^3/mm^3
  Baseline (n= 20, 20, 21) | 81.75 (58.39) | 68.50 (30.40) | 75.67 (38.96)
  Day 14 (n= 18, 19, 18) | 93.06 (50.13) | 109.47 (73.60) | 81.61 (39.43)
  Month 1 (n= 19, 18, 19) | 94.37 (31.58) | 87.39 (33.55) | 101.37 (50.30)
  Month 3 (n= 19, 17, 20) | 83.00 (41.52) | 90.94 (31.64) | 85.90 (30.19)
  Month 6 (n= 16, 14, 18) | 79.81 (43.02) | 73.07 (12.46) | 71.89 (30.85)

15. Secondary Outcome: Trough Levels of Tacrolimus (TAC)
Time Frame: Pre-dose on Day 14, Month 1, 3, 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Tacrolimus
Number analyzed (Participants) | 18
nanogram/milliliter (ng/mL)
  Day 14 (n= 18) | 11.17 (4.15)
  Month 1 (n= 18) | 9.11 (3.20)
  Month 3 (n= 17) | 8.82 (4.05)
  Month 6 (n= 15) | 8.33 (4.06)

16. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36) Version 2.0 (V2)
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. These 8 aspects can also be summarized as physical and mental component scores (CS). Total of 11 variables were analyzed (8 subscales, 2 composite subscales and Question 2 "how would you rate your health in general now?" (range 1= better, 5= worst). The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Baseline, Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 16 | 17 | 17
units on a scale
  Bodily pain: Baseline (n= 16, 17, 17) | 49.89 (10.55) | 52.15 (10.91) | 50.46 (11.14)
  Bodily pain: Month 6 (n=15, 10, 17) | 54.79 (10.30) | 55.06 (8.77) | 57.54 (8.93)
  General health: Baseline (n= 15, 17, 17) | 44.48 (10.72) | 43.40 (9.47) | 43.65 (7.46)
  General health: Month 6 (n= 15, 10, 17) | 49.79 (8.12) | 49.50 (6.71) | 53.80 (8.85)
  Mental CS: Baseline (n= 15, 17, 17) | 45.18 (13.79) | 42.15 (12.20) | 46.73 (8.40)
  Mental CS: Month 6 (n= 15, 10, 17) | 52.38 (11.18) | 56.18 (5.22) | 51.62 (9.11)
  Mental health: Baseline (n= 16, 17, 17) | 47.90 (11.84) | 46.53 (10.79) | 49.68 (7.64)
  Mental health: Month 6 (n= 15, 10, 17) | 52.82 (11.16) | 54.51 (5.97) | 51.17 (8.45)
  Physical CS: Baseline (n= 15, 17, 17) | 45.37 (8.60) | 44.71 (10.76) | 41.11 (9.76)
  Physical CS: Month 6 (n= 15, 10, 17) | 50.67 (8.98) | 49.76 (6.31) | 53.87 (8.87)
  Physical functioning: Baseline (n= 16, 17, 17) | 47.30 (8.31) | 43.79 (12.69) | 41.20 (13.43)
  Physical functioning: Month 6 (n= 15, 10, 17) | 47.49 (12.03) | 48.40 (7.58) | 50.72 (10.28)
  Q2: Baseline (n= 16, 17, 17) | 3.25 (1.24) | 3.18 (1.33) | 2.59 (1.06)
  Q2: Month 6 (n= 15, 10, 17) | 1.07 (0.26) | 1.10 (0.32) | 1.41 (1.06)
  Role emotional: Baseline (n= 16, 17, 17) | 41.06 (17.34) | 37.81 (16.20) | 39.64 (15.26)
  Role emotional: Month 6 (n= 15, 10, 17) | 48.36 (12.51) | 52.77 (8.56) | 49.70 (13.33)
  Role physical: Baseline (n= 16, 17, 17) | 38.64 (12.74) | 36.69 (12.35) | 33.66 (8.84)
  Role physical: Month 6 (n= 15, 10, 17) | 51.14 (8.81) | 50.73 (9.25) | 50.51 (11.09)
  Social functioning: Baseline (n= 16, 17, 17) | 39.46 (13.24) | 41.45 (10.95) | 42.73 (10.75)
  Social functioning: Month 6 (n= 15, 10, 17) | 51.03 (8.36) | 53.58 (5.27) | 50.75 (9.62)
  Vitality: Baseline (n= 16, 17, 17) | 46.43 (12.55) | 43.46 (11.12) | 46.77 (9.29)
  Vitality: Month 6 (n= 15, 10, 17) | 56.25 (10.66) | 58.65 (4.76) | 58.52 (10.73)

17. Secondary Outcome: End-Stage Renal Disease Symptom Checklist-Transplantation Module (ESRD-SCL)
Description: ESRD-SCL:43-item disease specific self-administered questionnaire. Participants' rated question"At the moment,how much do you suffer?"for each item on 5 point scale,ranged (Ra) 0(not at all)to 4(extremely).Consisted of 6 subscales:cardiac and renal dysfunction;Ra 0-28,increased(In) growth of gum and hair;Ra 0-20,limited cognitive capacity;Ra 0-32,limited physical capacity;Ra 0-40,side effects (SEs) of corticosteroids;Ra 0-20,transplantation associated psychological distress(TAPD);Ra 0-32(higher scores=greater dysfunction for each subscale).Total score:0-172,higher scores=greater dysfunction.
Time Frame: Baseline, Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 15 | 15 | 17
units on a scale
  Cardiac and renal dysfunction:Baseline(n=13,15,17) | 0.60 (0.43) | 0.78 (0.68) | 0.67 (0.60)
  Cardiac and renal dysfunction:Month 6(n=15,10,16) | 0.26 (0.27) | 0.30 (0.32) | 0.22 (0.28)
  In growth of gum and hair: Baseline (n=14,15,17) | 0.19 (0.36) | 0.11 (0.15) | 0.13 (0.26)
  In growth of gum and hair: Month 6 (n=15,9,16) | 0.17 (0.27) | 0.11 (0.15) | 0.10 (0.22)
  Limited cognitive capacity: Baseline (n=14,15,17) | 0.68 (0.65) | 0.58 (0.69) | 0.78 (0.57)
  Limited cognitive capacity: Month 6 (n=15,10,17)) | 0.55 (0.49) | 0.16 (0.31) | 0.35 (0.46)
  Limited physical capacity: Baseline (n=14,15,17) | 0.65 (0.46) | 0.77 (0.57) | 0.62 (0.35)
  Limited physical capacity: Month 6 (n=15,10,16) | 0.41 (0.39) | 0.49 (0.48) | 0.38 (0.53)
  SEs of corticosteroids: Baseline (n=13,15,17) | 0.58 (0.64) | 0.44 (0.51) | 0.68 (0.74)
  SEs of corticosteroids: Month 6 (n=15,10,16) | 0.65 (0.78) | 0.52 (0.48) | 0.24 (0.43)
  TAPD: Baseline (n=14,15,17) | 1.10 (0.68) | 1.14 (0.78) | 0.97 (0.47)
  TAPD: Month 6 (n=15,10,16) | 0.69 (0.44) | 0.51 (0.36) | 0.58 (0.70)

18. Secondary Outcome: Healthcare Resource Utilization Questionnaire (HCRUQ)
Description: Healthcare Resource Utilization Questionnaire (HCRUQ) was used to assess healthcare resources which included number of events such as physician and other health professional visits, number of treatments or diagnostic tests, number of hospitalizations, and number of emergency room visits.
Time Frame: Baseline, Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: events
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 16 | 16 | 17
events
  Physician visits: Baseline (n= 15, 16, 17) | 3.33 (4.15) | 4.31 (4.74) | 4.47 (6.32)
  Physician visits: Month 6 (n= 10, 7, 10) | 4.20 (6.34) | 7.29 (8.88) | 8.70 (8.63)
  Emergency room visits: Baseline (n= 16, 16, 17) | 0.06 (0.25) | 0.19 (0.40) | 0.00 (0.00)
  Emergency room visits: Month 6 (n= 10, 7, 10) | 0.50 (0.85) | 0.14 (0.38) | 0.10 (0.32)
  Diagnostic tests: Baseline (n= 14, 16, 17) | 7.14 (8.56) | 5.88 (6.06) | 16.06 (28.45)
  Diagnostic tests: Month 6 (n= 10, 7, 10) | 0.40 (0.97) | 0.86 (1.21) | 4.20 (12.25)
  Hospital visits: Baseline (n= 15, 16, 17) | 0.07 (0.26) | 0.00 (0.00) | 0.00 (0.00)
  Hospital visits: Month 6 (n= 10, 7, 10) | 0.60 (1.07) | 0.43 (0.79) | 0.10 (0.32)

19. Secondary Outcome: Healthcare Resource Utilization Questionnaire (HCRUQ) - 5th Question
Description: Fifth question in the HCRUQ was "Upon discharge from the hospital, did you return to your previous place of residence?" and number of participants who responded "yes or no" to the question was reported.
Time Frame: Month 6
Population: FAS included all randomized participants who received at least 1 dose of study medication. Here, N (Number of participants analyzed) signifies participants evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 9 | 6 | 7
participants
  Yes | 7 | 6 | 6
  No | 2 | 0 | 1

20. Secondary Outcome: Glomerular Filtration Rate (GFR) by Cockcroft-Gault
Description: GFR: index of kidney function described the flow rate of filtered fluid through the kidney. GFR was measured directly or estimated using established formulas. GFR was calculated using Cockcroft-Gault equation. GFR by Cockcroft-Gault equation= body weight*(140 minus age in years) divided by (72*serum creatinine). For females, value obtained was multiplied by 0.85. A normal GFR is >90 mL/min, although children and older people usually have a lower GFR. Lower values indicated poor kidney function. A GFR <15 mL/min indicated kidney failure.
Time Frame: Day 14, Month 1, 3, 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 19 | 20
mL/min
  Day 14 (n= 19, 19, 20) | 73.24 (19.14) | 78.37 (20.08) | 76.14 (17.14)
  Month 1 (n= 20, 18, 19) | 80.73 (23.47) | 81.83 (11.54) | 79.90 (19.15)
  Month 3 (n= 18, 18, 20) | 81.84 (15.81) | 81.99 (14.95) | 86.86 (20.03)
  Month 6 (n= 17, 14, 18) | 82.17 (19.27) | 79.99 (19.72) | 91.89 (16.66)

21. Secondary Outcome: Glomerular Filtration Rate (GFR) by Modification of Diet in Renal Disease (MDRD) Equation
Description: GFR: index of kidney function described the flow rate of filtered fluid through the kidney. GFR was measured directly or estimated using established formulas. GFR was calculated using MDRD equation. GFR by MDRD equation= 170 * (serum creatinine) ^ (-0.999)*(age in years)^(-0.176)*(0.762 if female) * (1.18 if black)*(blood urea nitrogen concentration)^(-0.170)*(serum albumin concentration)^(0.318). Normal GFR is >90 mL/min/1.73 square meter (m^2), although children and older people usually have a lower GFR. Lower values indicated poor kidney function. A GFR <15 mL/min indicated kidney failure.
Time Frame: Day 14, Month 1, 3, 6
Population: FAS included all randomized participants who received at least 1 dose of study medication. Here, N (Number of participants analyzed) signifies participants evaluable for this measure and 'n' signifies those participants evaluable at specific time points for each group respectively.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 19 | 20
mL/min/1.73 m^2
  Day 14 (n= 19, 19, 20) | 60.67 (19.01) | 57.97 (16.32) | 56.70 (21.39)
  Month 1 (n= 20, 18, 19) | 66.82 (20.83) | 62.70 (9.50) | 62.55 (22.47)
  Month 3 (n= 18, 18, 20) | 64.58 (13.68) | 62.04 (12.46) | 66.45 (22.00)
  Month 6 (n= 17, 14, 18) | 63.59 (12.02) | 58.95 (16.19) | 68.29 (22.10)

22. Secondary Outcome: Glomerular Filtration Rate (GFR) by Reciprocal of Serum Creatinine (1/sCr)
Description: GFR is a measure of renal function. The reciprocal of serum creatinine is an estimate of GFR.
Time Frame: Day 14, Month 1, 3, 6
Population: FAS included all randomized participants who received at least 1 dose of study medication. Here, N (Number of participants analyzed) signifies participants evaluable for this measure and 'n' signifies those participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: deciliter/mg (dL/mg)
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 19 | 20
deciliter/mg (dL/mg)
  Day 14 (n= 19, 19, 20) | 0.87 (0.28) | 0.75 (0.19) | 0.75 (0.24)
  Month 1 (n= 20, 18, 19) | 0.91 (0.30) | 0.79 (0.14) | 0.78 (0.24)
  Month 3 (n= 18, 18, 20) | 0.86 (0.21) | 0.77 (0.18) | 0.82 (0.21)
  Month 6 (n= 17, 14, 18) | 0.86 (0.19) | 0.73 (0.19) | 0.84 (0.19)

23. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 2 months after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to Month 8 (2 months follow-up)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
participants
  AEs | 20 | 18 | 21
  SAEs | 8 | 10 | 6

24. Secondary Outcome: Number of Participants With First Clinically Significant Infection
Description: Clinically significant (Viral, Bacterial and Fungal) infection was defined as the presence of presumed or documented infection confirmed by culture, biopsy, genomic or serologic findings post-randomization and required hospitalization or anti-infective treatment, or otherwise deemed significant by the Investigator.
Time Frame: Month 3, 6
Population: FAS included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
participants
  Month 3 | 2 | 7 | 3
  Month 6 | 6 | 11 | 5

25. Secondary Outcome: Number of Participants With New Onset Diabetes Mellitus (NODM)
Time Frame: Month 3, 6
Population: FAS included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
participants
  Month 3 | 0 | 0 | 2
  Month 6 | 1 | 0 | 2

26. Secondary Outcome: Fasting Serum Glucose Levels
Time Frame: Baseline, Day 14, Month 1, 3, 6
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication. Here, N (Number of participants analyzed) signifies participants evaluable for this measure and 'n' signifies those participants evaluable at specific time points for each arm group respectively.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 19 | 21
mg/dL
  Baseline: (n= 18, 19, 21) | 114.50 (63.72) | 102.68 (63.26) | 90.29 (19.87)
  Day 14 (n= 19, 19, 20) | 131.58 (85.36) | 95.58 (32.45) | 99.85 (32.43)
  Month 1 (n= 20, 18, 19) | 120.35 (90.42) | 85.22 (18.40) | 99.16 (29.37)
  Month 3 (n= 18, 18, 20) | 93.56 (21.94) | 92.56 (34.75) | 101.05 (22.79)
  Month 6 (n= 17, 14, 18) | 108.76 (36.78) | 94.57 (19.41) | 95.11 (22.68)

27. Secondary Outcome: Number of Participants With Hypercholesterolemia
Description: Hypercholesterolemia is a condition characterized by very high levels of cholesterol in the blood. Hypercholesterolemia was defined as a value of total serum cholesterol greater than 240 mg/dL.
Time Frame: Baseline, Day 14, Month 1, 3, 6
Population: as for outcome 26
Measure: Number; unit: participants
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 19 | 21
participants
  Baseline (n= 18, 19, 21) | 1 | 1 | 0
  Day 14 (n= 19, 19, 20) | 5 | 5 | 1
  Month 1 (n= 20, 18, 19) | 8 | 6 | 2
  Month 3 (n= 18, 18, 20) | 5 | 5 | 2
  Month 6 (n= 17, 14, 18) | 4 | 3 | 1

28. Secondary Outcome: Total Serum Cholesterol, Low Density Lipoprotein (LDL) and High Density Lipoprotein (HDL) Levels
Time Frame: Baseline, Day 14, Month 1, 3, 6
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 19 | 21
mg/dL
  Total serum cholesterol: Baseline (n=18,19,21) | 168.78 (34.33) | 159.79 (39.20) | 166.86 (38.25)
  Total serum cholesterol: Day 14 (n=19,19,20) | 217.21 (44.79) | 208.05 (56.37) | 184.95 (36.79)
  Total serum cholesterol: Month 1 (n=20,18,19) | 245.20 (48.51) | 232.17 (66.17) | 202.89 (31.94)
  Total serum cholesterol: Month 3 (n=18,18,20) | 216.17 (38.92) | 203.00 (49.34) | 193.90 (39.74)
  Total serum cholesterol: Month 6 (n=17,14,18) | 207.88 (36.01) | 206.07 (38.72) | 195.50 (43.28)
  LDL: Baseline (n=18,18,19) | 93.17 (28.08) | 87.78 (27.85) | 90.74 (31.76)
  LDL: Day 14 (n=17,19,20) | 114.71 (36.60) | 113.05 (38.08) | 98.70 (25.81)
  LDL: Month 1 (n=18,18,19) | 139.28 (35.85) | 130.50 (48.80) | 110.32 (26.78)
  LDL: Month 3 (n=18,18,20) | 118.72 (33.15) | 114.06 (35.10) | 111.50 (34.87)
  LDL: Month 6 (n=17,14,18) | 117.00 (27.20) | 119.00 (28.21) | 114.50 (36.61)
  HDL: Baseline (n=18,19,21) | 43.89 (13.01) | 36.84 (12.76) | 46.00 (11.75)
  HDL: Day 14 (n=19,19,20) | 61.58 (13.20) | 64.16 (16.54) | 55.05 (16.77)
  HDL: Month 1 (n=20,18,19) | 75.65 (19.26) | 69.06 (21.29) | 62.16 (19.66)
  HDL: Month 3 (n=18,18,20) | 66.17 (16.51) | 56.11 (17.88) | 54.05 (13.80)
  HDL: Month 6 (n=17,14,18) | 59.53 (18.43) | 51.50 (12.78) | 55.00 (14.97)

29. Secondary Outcome: Number of Participants With Hypertriglyceridemia
Description: Hypertriglyceridemia was defined as a value of triglycerides greater than 200 mg/dL.
Time Frame: Baseline, Day 14, Month 1, 3, 6
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication. Here, N (Number of participants analyzed) signifies participants evaluable for this measure and 'n' signifies those participants evaluable at specific time points for each group respectively.
Measure: Number; unit: participants
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 19 | 21
participants
  Baseline (n= 18, 19, 21) | 4 | 7 | 5
  Day 14 (n= 19, 19, 20) | 7 | 2 | 6
  Month 1 (n= 20, 18, 19) | 7 | 5 | 3
  Month 3 (n= 18, 18, 20) | 5 | 5 | 2
  Month 6 (n= 17, 14, 18) | 5 | 5 | 1

30. Secondary Outcome: Supine Systolic and Diastolic Blood Pressure (BP)
Time Frame: Baseline, Day 2, 3, 14, Month 1, 3, 6
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication. Here 'n' signifies those participants evaluable at specific time points for each arm group respectively.
Measure: Mean (Standard Deviation); unit: millimeter of mercury
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
millimeter of mercury
  Diastolic BP (DBP) : Baseline (n= 20, 20, 21) | 77.10 (14.04) | 75.25 (9.95) | 76.52 (17.71)
  DBP: Day 2 (n= 19, 20, 20) | 79.05 (13.62) | 80.20 (9.68) | 78.50 (10.37)
  DBP: Day 3 (n= 18, 19, 18) | 82.50 (10.59) | 88.05 (9.45) | 82.61 (9.67)
  DBP: Day 14 (n= 20, 19, 20) | 78.45 (11.83) | 81.21 (8.15) | 75.20 (7.29)
  DBP: Month 1 (n= 20, 18, 19) | 78.95 (11.08) | 80.83 (9.29) | 76.32 (11.61)
  DBP: Month 3 (n= 19, 18, 21) | 80.42 (10.91) | 76.06 (12.66) | 77.33 (10.88)
  DBP: Month 6 (n= 17, 13, 19) | 77.24 (10.46) | 83.23 (10.21) | 79.00 (9.99)
  Systolic BP (SBP): Baseline (n= 20, 20, 21) | 139.65 (23.22) | 139.45 (18.98) | 136.24 (27.68)
  SBP: Day 2 (n= 19, 20, 20) | 141.16 (18.66) | 143.55 (13.87) | 136.05 (20.14)
  SBP: Day 3 (n= 18, 19, 18) | 146.78 (17.33) | 152.42 (14.47) | 139.94 (18.13)
  SBP: Day 14 (n= 20, 19, 20) | 135.90 (24.43) | 141.16 (19.48) | 121.45 (17.01)
  SBP: Month 1 (n= 20, 18, 19) | 129.05 (19.06) | 136.22 (15.01) | 128.21 (13.57)
  SBP: Month 3 (n= 19, 18, 21) | 140.32 (20.58) | 133.44 (20.05) | 124.00 (14.65)
  SBP: Month 6 (n= 17, 13, 19) | 135.76 (17.08) | 134.31 (14.82) | 128.00 (17.94)

31. Secondary Outcome: Number of Participants With Drug Usage
Description: Lipid lowering agents, antihypertensive agents, oral hypoglycemic agents (OHA) , anti-diabetic agents (ADA) and insulin drug usage was collected.
Time Frame: Baseline, Day 14, Month 1, 3, 6
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
participants
  Lipid Lowering: Baseline ( n= 20, 20, 21) | 6 | 9 | 9
  Lipid Lowering: Day 14 (n= 20, 19, 21) | 3 | 4 | 4
  Lipid Lowering: Month 1 (n= 20, 19, 21) | 5 | 5 | 4
  Lipid Lowering: Month 3 (n= 20, 19, 20) | 8 | 9 | 5
  Lipid Lowering: Month 6 (n= 18, 15, 20) | 10 | 8 | 7
  Antihypertensive: Baseline ( n= 20, 20, 21) | 17 | 18 | 18
  Antihypertensive: Day 14 (n= 20, 19, 21) | 15 | 19 | 15
  Antihypertensive: Month 1 (n= 20, 19, 21) | 15 | 18 | 16
  Antihypertensive: Month 3 (n= 20, 19, 20) | 16 | 18 | 17
  Antihypertensive: Month 6 (n= 18, 15, 20) | 14 | 11 | 16
  OHA, ADA, insulin usage: Baseline (n= 20, 20, 21) | 9 | 7 | 5
  OHA, ADA, insulin usage: Day 14 (n= 20, 19, 21) | 5 | 4 | 3
  OHA, ADA, insulin usage: Month 1 (n= 20, 19, 21) | 5 | 4 | 3
  OHA, ADA, insulin usage: Month 3 (n= 20, 19, 20) | 5 | 4 | 3
  OHA, ADA, insulin usage: Month 6 (n= 18, 15, 20) | 6 | 3 | 2

32. Secondary Outcome: Epstein Barr Virus (EBV) and Cytomegalovirus (CMV) Deoxyribonucleic Acid (DNA) Load
Time Frame: Baseline, Month 1, 3, 6 for CMV; Baseline, Day 14, Month 1, 3, 6 for EBV
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Copies/500 ng DNA
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 19 | 20
Copies/500 ng DNA
  EBV: Baseline (n= 20, 19, 19) | 2.65 (11.39) | 0.26 (0.81) | 3.21 (11.27)
  EBV: Day 14 (n= 18, 19, 20) | 4.22 (13.82) | 0.58 (0.90) | 3.60 (9.32)
  EBV: Month 1 (n= 20, 18, 18) | 5.25 (20.97) | 0.50 (0.92) | 1.94 (5.23)
  EBV: Month 3 (n= 18, 18, 20) | 0.28 (0.57) | 0.28 (0.46) | 0.65 (1.95)
  EBV: Month 6 (n= 15, 13, 18) | 0.73 (1.79) | 15.15 (27.62) | 0.61 (1.46)
  CMV: Baseline (n= 20, 19, 19) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  CMV: Month 1 (n= 20, 18, 18) | 0.15 (0.49) | 43.50 (184.55) | 0.00 (0.00)
  CMV: Month 3 (n= 18, 18, 20) | 55.67 (235.67) | 4.06 (16.71) | 0.05 (0.22)
  CMV: Month 6 (n= 15, 13, 18) | 58.87 (226.33) | 2.38 (5.45) | 0.00 (0.00)

33. Secondary Outcome: BK Virus (BKV) Deoxyribonucleic Acid (DNA) Load
Time Frame: Baseline, Month 1, 3, 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Copies/20 mcL plasma
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 19 | 20
Copies/20 mcL plasma
  Baseline (n= 20, 19, 19) | 0.00 (0.00) | 0.05 (0.23) | 0.05 (0.23)
  Month 1 (n= 20, 18, 18) | 0.00 (0.00) | 5.33 (22.13) | 0.00 (0.00)
  Month 3 (n= 18, 18, 20) | 0.00 (0.00) | 7.56 (21.55) | 7.95 (28.96)
  Month 6 (n= 15, 13, 18) | 5.07 (16.55) | 189.85 (664.27) | 0.06 (0.24)

34. Secondary Outcome: Number of Participants With Cytomegalovirus (CMV) Disease
Time Frame: Month 3, 6
Population: FAS included all randomized participants who received at least 1 dose of study medication and based on time due to lost of follow-up, or up to Month 6. Here, N (Number of participants analyzed) signifies participants evaluable for this measure and 'n' signifies those participants evaluable at specific time points for each arm group respectively.
Measure: Number; unit: participants
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 19 | 20
participants
  Month 3 (n= 20, 19, 20) | 0 | 4 | 0
  Month 6 (n= 19, 16, 20) | 2 | 4 | 0

35. Secondary Outcome: Total White Blood Cells (WBC), Absolute Basophil, Absolute Eosinophil, Absolute Lymphocyte, Absolute Monocyte, Absolute Neutrophil
Time Frame: Baseline, Day 14, Month 1, 3, 6
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication. Here 'n' signifies those participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: cells*10^3/mm^3
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
cells*10^3/mm^3
  WBC: Baseline (n= 20, 20, 21) | 12.75 (3.79) | 11.09 (3.57) | 11.82 (5.16)
  WBC: Day 14 (n= 18, 19, 18) | 12.76 (3.68) | 13.81 (3.49) | 10.24 (3.10)
  WBC: Month 1 (n= 19,18, 19) | 7.33 (1.85) | 7.41 (2.80) | 7.43 (2.08)
  WBC: Month 3 (n= 19, 17, 20) | 5.47 (2.52) | 6.15 (2.82) | 5.48 (1.85)
  WBC: Month 6 (n= 16, 14, 18) | 5.57 (1.95) | 5.11 (2.22) | 6.06 (2.89)
  Basophil: Baseline (n= 20, 20, 21) | 0.04 (0.05) | 0.01 (0.03) | 0.02 (0.04)
  Basophil: Day 14 (n= 18, 19, 18) | 0.09 (0.07) | 0.11 (0.08) | 0.05 (0.05)
  Basophil: Month 1 (n= 19,18, 19) | 0.05 (0.08) | 0.07 (0.06) | 0.06 (0.05)
  Basophil: Month 3 (n= 19, 17, 20) | 0.04 (0.05) | 0.05 (0.05) | 0.04 (0.05)
  Basophil: Month 6 (n= 16, 14, 18) | 0.04 (0.05) | 0.04 (0.05) | 0.06 (0.06)
  Eosinophil: Baseline (n= 20, 20, 21) | 0.08 (0.08) | 0.06 (0.08) | 0.12 (0.20)
  Eosinophil: Day 14 (n= 18, 19, 18) | 0.17 (0.13) | 0.21 (0.12) | 0.13 (0.08)
  Eosinophil: Month 1 (n= 19,18, 19) | 0.14 (0.10) | 0.19 (0.16) | 0.13 (0.09)
  Eosinophil: Month 3 (n= 19, 17, 20) | 0.10 (0.03) | 0.11 (0.07) | 0.11 (0.07)
  Eosinophil: Month 6 (n= 16, 14, 18) | 0.11 (0.05) | 0.11 (0.08) | 0.17 (0.12)
  Lymphocyte: Baseline (n= 20, 20, 21) | 0.61 (0.41) | 0.52 (0.23) | 0.75 (0.45)
  Lymphocyte: Day 14 (n= 18, 19, 18) | 2.03 (1.43) | 2.48 (1.40) | 1.84 (0.93)
  Lymphocyte: Month 1 (n= 19,18, 19) | 1.96 (1.22) | 1.77 (0.79) | 1.81 (0.76)
  Lymphocyte: Month 3 (n= 19, 17, 20) | 1.26 (0.57) | 1.61 (0.97) | 1.29 (0.56)
  Lymphocyte: Month 6 (n= 16, 14, 18) | 1.44 (0.61) | 1.28 (0.81) | 1.47 (0.68)
  Monocyte: Baseline (n= 20, 20, 21) | 0.58 (0.44) | 0.39 (0.22) | 0.44 (0.26)
  Monocyte: Day 14 (n= 18, 19, 18) | 0.36 (0.16) | 0.41 (0.19) | 0.34 (0.14)
  Monocyte: Month 1 (n= 19,18, 19) | 0.26 (0.12) | 0.32 (0.13) | 0.28 (0.09)
  Monocyte: Month 3 (n= 19, 17, 20) | 0.31 (0.17) | 0.34 (0.19) | 0.28 (0.09)
  Monocyte: Month 6 (n= 16, 14, 18) | 0.31 (0.15) | 0.25 (0.15) | 0.34 (0.12)
  Neutrophil: Baseline (n= 20, 20, 21) | 11.63 (3.73) | 10.06 (3.53) | 10.37 (4.84)
  Neutrophil: Day 14 (n= 18, 19, 18) | 10.01 (3.14) | 10.48 (3.05) | 7.78 (2.99)
  Neutrophil: Month 1 (n= 19,18, 19) | 4.85 (1.86) | 4.93 (2.50) | 5.05 (1.82)
  Neutrophil: Month 3 (n= 19, 17, 20) | 3.68 (2.21) | 3.96 (2.01) | 3.72 (1.90)
  Neutrophil: Month 6 (n= 16, 14, 18) | 3.68 (1.67) | 3.37 (1.65) | 3.94 (2.27)

36. Secondary Outcome: Absolute Platelet Levels
Time Frame: Baseline, Day 14, Month 1, 3, 6
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: platelets*10^3/mm^3
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
platelets*10^3/mm^3
  Platelet: Baseline (n= 20, 20, 21) | 186.75 (59.33) | 204.85 (54.44) | 195.19 (47.97)
  Platelet: Day 14 (n= 18, 19, 18) | 330.17 (107.04) | 367.84 (101.31) | 301.28 (90.95)
  Platelet: Month 1 (n= 19,18, 19) | 249.68 (73.70) | 274.50 (88.30) | 276.79 (72.08)
  Platelet: Month 3 (n= 19, 17, 20) | 273.84 (89.95) | 307.00 (92.40) | 241.60 (66.80)
  Platelet: Month 6 (n= 16, 14, 18) | 272.19 (88.19) | 263.43 (109.78) | 225.17 (59.53)

37. Secondary Outcome: Hemoglobin Level
Description: Hemoglobin is the protein molecule in red blood cells that carries oxygen from the lungs to the body's tissues and returns carbon dioxide from the tissues back to the lungs.
Time Frame: Baseline, Day 14, Month 1, 3, 6
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
g/dL
  Baseline (n= 20, 20, 21) | 11.04 (1.48) | 10.65 (1.43) | 11.84 (1.37)
  Day 14 (n= 19, 19, 18) | 11.83 (1.29) | 11.68 (0.89) | 11.93 (1.67)
  Month 1 (n= 19, 18, 19) | 12.16 (1.04) | 12.29 (1.12) | 12.20 (1.42)
  Month 3 (n= 19, 17, 20) | 12.35 (1.79) | 12.20 (1.55) | 12.91 (1.43)
  Month 6 (n= 16, 14, 18) | 12.83 (1.54) | 12.41 (1.99) | 14.26 (1.32)

38. Secondary Outcome: Hematocrit Level
Description: The hematocrit is recorded as the percentage of volume of red blood cells (RBCs) in a blood sample.
Time Frame: Baseline, Day 14, Month 1, 3, 6
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: percentage of blood
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
percentage of blood
  Baseline (n= 20, 20, 21) | 34.75 (4.82) | 33.30 (5.02) | 36.86 (5.18)
  Day 14 (n= 18, 19, 18) | 37.78 (3.73) | 37.16 (3.50) | 37.11 (4.83)
  Month 1 (n= 19, 18, 19) | 38.74 (2.81) | 38.22 (3.89) | 37.95 (3.99)
  Month 3 (n= 19, 17, 20) | 38.53 (5.30) | 37.12 (4.37) | 39.50 (4.05)
  Month 6 (n= 16, 14, 18) | 40.19 (3.75) | 37.86 (6.14) | 43.67 (3.88)

39. Secondary Outcome: Alanine Aminotransferase (ALT) Level
Description: ALT is the enzyme found in the liver and it is measured to see if the liver is damaged or diseased.
Time Frame: Baseline, Day 14, Month 1, 3, 6
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication. Here, 'n' signifies those participants evaluable at specific time points for each arm group respectively.
Measure: Mean (Standard Deviation); unit: unit/liter
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
unit/liter
  Baseline (n= 19, 20, 21) | 24.84 (18.52) | 18.45 (9.39) | 18.33 (10.36)
  Day 14 (n= 19, 19, 20) | 39.05 (35.77) | 70.63 (66.72) | 31.50 (27.89)
  Month 1 (n= 20, 18, 19) | 28.95 (14.16) | 56.39 (57.47) | 21.32 (10.72)
  Month 3 (n= 18, 18, 20) | 26.28 (10.56) | 36.22 (31.40) | 16.10 (6.98)
  Month 6 (n= 17, 14, 18) | 31.06 (20.31) | 37.86 (19.81) | 23.28 (21.50)

40. Secondary Outcome: Electrocardiogram (ECG) Parameters
Description: ECG parameters included PR interval, QT interval, corrected QT using Bazett's formula (QTcB) and QTc using Fridericia's formula (QTcF) interval, and QRS width.
Time Frame: Baseline, Month 3, 6
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 19 | 16 | 19
millisecond
  PR: Baseline (n= 15, 11, 17) | 147.60 (21.18) | 141.82 (50.77) | 151.53 (16.92)
  PR: Month 3 (n= 19, 15, 18) | 156.37 (20.22) | 156.00 (59.08) | 150.17 (20.38)
  PR: Month 6 (n= 16, 13, 19) | 161.44 (24.43) | 163.23 (26.94) | 154.53 (23.21)
  QT: Baseline (n= 15, 12, 17) | 412.40 (38.35) | 404.50 (43.33) | 393.88 (34.75)
  QT: Month 3 (n= 19, 16, 18) | 383.32 (38.00) | 378.88 (28.47) | 384.00 (33.23)
  QT: Month 6 (n= 16, 13, 19) | 401.44 (28.53) | 383.85 (33.68) | 384.68 (20.24)
  QTcB: Baseline (n= 15, 12, 17) | 454.77 (27.29) | 447.37 (36.95) | 447.42 (22.44)
  QTcB: Month 3 (n= 19, 16, 18) | 417.25 (27.22) | 412.23 (29.22) | 409.81 (34.15)
  QTcB: Month 6 (n= 16, 13, 19) | 416.83 (21.01) | 410.48 (22.24) | 413.55 (25.05)
  QTcF: Baseline (n= 15, 12, 17) | 439.77 (25.54) | 432.22 (34.93) | 428.57 (23.95)
  QTcF: Month 3 (n= 19, 16, 18) | 405.05 (23.63) | 400.60 (25.74) | 400.62 (28.63)
  QTcF: Month 6 (n= 16, 13, 19) | 411.44 (20.17) | 401.24 (24.06) | 403.41 (17.51)
  QRS: Baseline (n= 15, 12, 17) | 88.80 (12.21) | 102.67 (29.47) | 92.82 (9.08)
  QRS: Month 3 (n= 19, 16, 18) | 87.74 (14.18) | 102.13 (39.78) | 88.22 (10.14)
  QRS: Month 6 (n= 16, 13, 19) | 91.75 (16.13) | 90.31 (32.15) | 89.74 (9.89)

41. Secondary Outcome: Number of Participants With Discontinuation
Time Frame: Month 1, 2, 3, 4, 5, 6
Population: FAS included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Number analyzed (Participants) | 20 | 20 | 21
participants
  Month 1 | 0 | 1 | 0
  Month 2 | 1 | 1 | 0
  Month 3 | 1 | 1 | 1
  Month 4 | 1 | 2 | 1
  Month 5 | 2 | 4 | 1
  Month 6 | 2 | 6 | 1

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-690,550 15 mg | CP-690,550 30 mg | Tacrolimus
Serious Adverse Events (participants affected / at risk) | 8/20 | 10/20 | 6/21
Other Adverse Events (participants affected / at risk) | 20/20 | 18/20 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 15 mg (N=20) | CP-690,550 30 mg (N=20) | Tacrolimus (N=21)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 2 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Kidney transplant rejection (Immune system disorders) | 1 | 2 | 0
Transplant rejection (Immune system disorders) | 1 | 2 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 0
BK virus infection (Infections and infestations) | 0 | 2 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 2 | 3 | 0
Endocarditis bacterial (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ureteric injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 2 | 1
Blood glucose abnormal (Investigations) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0 | 0
Lupus nephritis (Renal and urinary disorders) | 0 | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 15 mg (N=20) | CP-690,550 30 mg (N=20) | Tacrolimus (N=21)
Anaemia (Blood and lymphatic system disorders) | 5 | 6 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 2 | 4
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocythaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 2 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 0
Anal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 6 | 5
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 5
Dyspepsia (Gastrointestinal disorders) | 3 | 4 | 2
Erosive duodenitis (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 3
Asthenia (General disorders) | 0 | 1 | 1
Catheter site pain (General disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 1
Chills (General disorders) | 2 | 0 | 0
Fatigue (General disorders) | 3 | 2 | 0
Feeling jittery (General disorders) | 0 | 0 | 1
Irritability (General disorders) | 0 | 1 | 1
Oedema (General disorders) | 1 | 1 | 0
Oedema peripheral (General disorders) | 4 | 5 | 7
Pain (General disorders) | 1 | 0 | 2
Pitting oedema (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 4 | 1
Swelling (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Kidney transplant rejection (Immune system disorders) | 0 | 0 | 1
BK virus infection (Infections and infestations) | 0 | 1 | 0
Candidiasis (Infections and infestations) | 0 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0
Human polyomavirus infection (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Tinea versicolour (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 5 | 2
Wound infection (Infections and infestations) | 0 | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incision site complication (Injury, poisoning and procedural complications) | 2 | 3 | 1
Incision site pain (Injury, poisoning and procedural complications) | 3 | 0 | 2
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Medical device complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Medical device pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Open wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 4 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 2
Blood creatinine increased (Investigations) | 1 | 5 | 1
Blood testosterone decreased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Heart rate irregular (Investigations) | 1 | 0 | 0
Immunosuppressant drug level increased (Investigations) | 1 | 0 | 0
Vascular resistance systemic increased (Investigations) | 1 | 0 | 0
Viral test positive (Investigations) | 0 | 0 | 1
Virus urine test positive (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1
Weight increased (Investigations) | 0 | 2 | 2
White blood cell count increased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 3 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Aura (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 5
Headache (Nervous system disorders) | 3 | 2 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 2 | 0 | 9
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 2 | 5
Mood altered (Psychiatric disorders) | 0 | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 2 | 1
Haematuria (Renal and urinary disorders) | 2 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 3 | 1
Nephritis interstitial (Renal and urinary disorders) | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 2 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0
Oedema genital (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasopharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 5 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Medical device implantation (Surgical and medical procedures) | 0 | 1 | 0
Wound drainage (Surgical and medical procedures) | 1 | 0 | 1
Hot flush (Vascular disorders) | 0 | 2 | 0
Hypertension (Vascular disorders) | 3 | 5 | 2
Hypotension (Vascular disorders) | 1 | 0 | 0
Lymphocele (Vascular disorders) | 1 | 2 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Results for first BPAR, BPCAN, treatment and efficacy failure, rejection, clinically significant infections, NODM and discontinuation reported as number and not percentage as planned. Stage 2 of study was not conducted due to administrative reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.